CLINICAL TRIAL: NCT03657706
Title: Analysis of the Aesthetic Outcome After Root Coverage Using Tunneling Technique With Subepithelial Connective Tissue Graft Versus Tunneling Technique With Modified Free Gingival Graft in Miller's Class III Recession Defect: a Randomized Clinical Trial
Brief Title: Tunneling Technique in Treatment of Miller's Class III Gingival Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Abdallah Abdelkhalek, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-06-34
Record Dates: First submitted 2018-06-26; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — N-(N-(4-deoxy-4-amino-10-methylpteroyl)-4-fluoroglutamyl)-gamma-glutamate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): tunnel procedure with subepithelial connective tissue graft (sCTG)
  Interventions: Procedure: group A (Tunnel procedure with subepithelial connective tissue graft (sCTG)
- group B (Active Comparator): tunnel procedure with modified free gingival graft (mFGG)
  Interventions: Procedure: group B (Tunnel procedure with modified free gingival graft (mFGG))

INTERVENTIONS:
Procedure: group A (Tunnel procedure with subepithelial connective tissue graft (sCTG) — Subepithelial connective tissue graft (autogenous graft) will be harvested from the palate by Single incision technique to be used with the prepared tunnel to treating gingival recession
  Other Names: Tunnel procedure with subepithelial connective tissue graft (sCTG); Autogenous sCTG will be used with tunnel procedure
  Arms: group A
Procedure: group B (Tunnel procedure with modified free gingival graft (mFGG)) — modified free gingival graft (autogenous graft) will be harvested from the palate and will be used with the prepared tunnel to be used in treating gingival recession
  Other Names: Tunnel procedure with modified free gingival graft (mFGG); Autogenous mFGG will be used with tunnel procedure
  Arms: group B

SUMMARY:
Several surgical techniques have been proposed to correct recession defect and attain root coverage. Though, the majority were executed on Miller Class I and II recession defects. Moreover, Analysis of literature revealed only a few studies that treated miller class III recession defects.

In the current study, a new modification in the free gingival graft is proposed to provide the patient with more esthetic outcome, less pain and postoperative trauma. Likewise, the proposed graft modification will combined both FGG and CTG benefits, overcome the limitations of the FGG and enhances the advantages of CTG.

DETAILED DESCRIPTION:
In the current study, patients with Miller's class III will be randomly allocated in two groups. In the first group, gingival recession will be treated by tunneling technique with subepithelial connective tissue graft (sCTG). the tunnel preparation will be performed in the recession site then the sCTG will be harvested from the palate and inserted in the prepared tunnel and sutured in a coronally advanced position.

Equally , the second group will be treated with modified free gingival graft (mFGG). Initially, after tunnel preparation in the recession site and harvesting of the free gingival graft,the proposed modification is performed by mimicking the recession defect shape and size leaving the rest of the free gingival graft deepithelialized and inserted in the prepared tunnel. then, suturing will be performed in a coronally advanced position.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy systemic condition.
2. Buccal recession defects classified as Miller class III.
3. Clinical indication and/or patient request for recession coverage.
4. O'Leary index less than 20%.

Exclusion Criteria:

1. Pregnant females.
2. Smokers as smoking is a contraindication for any plastic periodontal surgery.
3. Unmotivated, uncooperative patients with poor oral hygiene
4. Patients with habits that may compromise the longevity and affect the result of the study as alcoholism or para-functional habits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
root coverage aesthetic score (RES) | 6 months
  RES evaluated five variables 6 months: gingival margin (GM), marginal tissue contour (MTC), soft tissue texture (STT), MGJ alignment, and gingival color (GC). Zero, 3, or 6 points were used for the evaluation of the position of the gingival margin, whereas a score of 0 or 1 point was used for each of the other variables.
  The ideal esthetic score was 10. Zero points were assigned if the final position of the gingival margin was equal or apical to the previous recession depth (failure of root coverage procedure), irrespective of color, the presence of a scar, MTC, or MGJ. Zero points were also assigned when a partial or total loss of interproximal papilla (black triangle) occurred following the treatment

SECONDARY OUTCOMES:
recession depth | 6 months
  Measured from the cemento-enamel junction the most apical extension of the gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
all the study records may be shared except that include participant name or personal information identifiers